CLINICAL TRIAL: NCT05388799
Title: The Effect of Brochure-Based Education on Surgical Fear and Anxiety in Patients Planned for Nose Surgery
Brief Title: The Effect of Brochure-Based Education on Patients Planned for Nose Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Sevgi Deniz Dogan, lecturer Dr., Cukurova University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 312256940
Record Dates: First submitted 2022-05-17; First posted 2022-05-24 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Nursing Caries
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- application group (Experimental): Before the operation, training will be given in line with the training brochure prepared by the researcher in the outpatient clinic and the printed version of the training brochure will be given to the patient. The training will be repeated by calling the patients the day before the surgery.
  Interventions: Other: Educational intervention
- control group (No Intervention): Standard care will be applied.

INTERVENTIONS:
Other: Educational intervention — In addition to standard care, brochure-supported education will be given to patients who are scheduled for nose surgery.
  Arms: application group

SUMMARY:
The study was planned as a randomized controlled trial to determine the effect of brochure-based education on fear and anxiety in patients scheduled for nose surgery.It is planned to collect research data in Hatay Mustafa Kemal University Hospital otorhinolaryngology clinic between June 2022 and June 2023.The population of the research will be the patients who are hospitalized in the otorhinolaryngology clinic of the aforementioned hospital and are planned for nasal surgery. The sample of the study, on the other hand, will consist of 52 patients who meet the inclusion criteria and agree to participate in the study verbally and in writing.The data of the study were collected by using the Personal Information Form, the Surgical Fear Scale and the Surgical Anxiety Scale, which were prepared in line with the literature.The data will be analyzed with the SPSS package program.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over, 65 years and under,
* Being literate,
* To be able to understand and speak Turkish
* First time nose surgery,
* Agreeing to participate in the research.

Exclusion Criteria:

* Having any psychiatric disorder that may reduce the ability to comprehend and understand
* The surgery was canceled for some reason.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
The effect of preoperative care on surgical fear in patients scheduled for nasal surgery | six months
  It will be evaluated with the 8-item Surgical Fear Scale, which was adapted into Turkish by Bağdigen and Karaman Özlü in 2016.It will be evaluated in the outpatient clinic before the surgery and in the clinic on the morning of the surgery.The score obtained from the items of the scale ranges from 0 to 10 (0 "I am not afraid at all", 10 "I am very afraid").The lowest score that can be obtained from the scale is 0, while the highest score is 80.The higher the score, the higher the patient's fear of surgery.
The effect of preoperative care on surgical anxiety in patients scheduled for nasal surgery | six months
  It will be evaluated with the 17-item Surgical Anxiety Scale adapted into Turkish by Göl and Bölükbaş.It will be evaluated in the outpatient clinic before the surgery and in the clinic on the morning of the surgery. The scale is in a five-point Likert type, scored as "never-0", "very little-1", "moderately-2", "very-3" and "extremely-4". The lowest score that can be obtained from the scale is 0, and the highest score is 68, and the higher the score, the higher the level of surgical anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Hatay Mustafa Kemal University Institute of Health Sciences, Hatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No